CLINICAL TRIAL: NCT05815654
Title: Research and Development of Warm Palace Analgesic Point Stickers Based on the Modern Technology of Traditional Chinese Medicine: Study Protocol for a Randomized Controlled Trial
Brief Title: Research and Development of WPAPS Based on the Modern Technology of Traditional Chinese Medicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Innovation and Technology Commission, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHX/004/20
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-10

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: 200 participants will be divided into experimental group and control group.
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly assigned to the experimental group (EG), or the placebo control group (CG) at a ratio of 5:5 stratified by recruitment site. Stratified block randomization will be used according to probability theory. An independent statistician will generate random sequences using R software version 4.2.1 (R Project for Statistical Computing, Vienna, Austria), in which the TCM syndrome type, duration, and the severity of dysmenorrhea will be used as indicators, after a patient's qualification is confirmed, a randomization number and its corresponding sticker will be provided to the assistant by the PI. Then the assistant will give the specific sticker to the subjects to ensure that both the assistant and the subjects will not know which type of sticker they get.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Palace Analgesic Point Sticker Group (Experimental): Participants in the EG group will be provided test sticker, containing Ding Xiang, Rou Gui, Gan Jiang, Huang Jie Zi, Rou Cong Rong, Xiao Hui Xiang, Hua Jiao, Ai Ye, Xiang Fu, Wu Zhu Yu, Graphene（0.01%）The acupoints for applying the sticker are Guanyuan (CV4), Zigong (EX-CA1), and Sanyinjiao (SP6). The subjects will be reminded to closely observe their skin during the process and remove the sticker in time if the subjects feel itchy or painful, and record the adverse event.
  Interventions: Device: Warm Palace Analgesic Point Sticker
- Control Group (Placebo Comparator): Participants in the CG group will be provided control sticker containing flour.The acupoints for applying the sticker are the same with experimental group
  Interventions: Device: Warm Palace Analgesic Point Sticker

INTERVENTIONS:
Device: Warm Palace Analgesic Point Sticker — The Warm Palace Analgesic Point Sticker is developed by Changchun University of Traditional Chinese Medicine

SUMMARY:
The goal of this double-blind randomized controlled trial is to determine the efficacy of Warm Palace Analgesic Point Sticker in relieving dysmenorrhea compared to placebo sticker. The main questions it aims to answer are:

* Can this Warm Palace Analgesic Point Sticker relieve dysmenorrhea?
* It is more effective to certain type of TCM syndrome differentiation? Qi stagnation and blood stasis syndrome or cold dampness syndrome?

Participants will :

* receive test sticker or control sticker five days before every menstruation, once a day, five hours each time, for five consecutive days
* take pictures of tongue
* fill in some questionnaires after treatment

DETAILED DESCRIPTION:
This study aims to determine the efficacy of Warm Palace Analgesic Point Sticker in relieving dysmenorrhea compared to placebo sticker through a double-blind, randomized controlled trial.

Two hundred participants will be enrolled. This trial consisting of an intervention phase for three menstrual cycles. After receiving an explanation of the trial and providing online informed consent, participants will be given screening numbers by registration order. Pain intensity of participants who completed the screening test will be assessed as baseline information during a run-in period. The run-in period will not exceed 40days. Before the run-in period, the participants will be offered an online diary and educated on how to record pain intensity using the Numerical Rating Scale (NRS) from one day before menstruation starts until menstruation ends. The participants will be forbidden to self-administer the medications presented in the exclusion or drop-out criteria. Participants with moderate or severe level of pain, average NRS pain scores greater than 4 on the first and second days of menstruation will be selected for enrollment in this trial, and the selected participants will receive randomly generated enrollment numbers. After the screening, the subjects will attend an online interview for evaluation, briefing, and tongue photo capturing and photo taking training. Then subjects will be randomly divided into two groups, the test sticker group, and the control sticker group. The total study period for each subject will be three months. Within three days from the end of the previous menstruation cycle, the participants will contact the research assistant, return their online diary, answer questionnaires regarding outcome measurements, and send back their tongue picture at each assessment. The intervention will be done during three menstrual cycles. One menstrual cycle may range from 21 to 40 days. We plan to conduct this trial for two years, starting from November 2022.

ELIGIBILITY:
Inclusion Criteria:

(1)18-35 years old; (2) Have a regular history of the menstrual cycle (28 days ± 7 days); (3) The first dysmenorrhea occurs before the age of 25, and at least 2 cycles after menarche; (4) No pregnancy/abortion / ectopic pregnancy history before the first dysmenorrhea; (5) Moderate to severe menstrual pain experienced at least 3 menstrual cycles prior to enrollment; (6) TCM syndrome differentiation is Qi stagnation and blood stasis syndrome and cold dampness syndrome.

Exclusion Criteria:

Women with secondary dysmenorrhea (include but not limited to endometriosis, pelvic inflammation or hysteromyoma) confirmed by gynaecologists through B-mode ultrasound; (2) Women with irregular menstrual cycle (menstruation is advanced or delayed no more than 7 days); (3) women who are suffering from uncontrollable nervous system diseases, immune deficiency, haemorrhagic diseases or other serious chronic diseases; (4) women who have taken prostaglandin synthase inhibitor (PGSI) two weeks before enrolment; (5) women who are lactating, pregnant or planning to pregnant in the next 6 months; (6) women who are taking drugs that may affect the results of the study (include but not limited to NSAIDs and oral contraceptives); (7) Women who are receiving moxibustion or have received moxibustion 2 weeks before enrolment; (8) Women who are participating in other clinical studies; (9) Those who cannot cooperate with application treatment; (10) Have a history of severe skin allergy and are allergic to more than 2 kinds of food or drugs.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Dysmenorrhea only occur to female.
Enrollment: 200 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Scores on the Cox Menstrual Symptom Scale at 3 Months | through study completion, an average of 3 months
  This scale was developed by the University of Virginia to evaluate the severity and duration of dysmenorrhea symptoms. The scale includes 17 items, all of which adopt the 5-level scoring method, in which 0 is for not noticeable / did not occur, 1 is for slightly bothersome / lasted less than 3 hours, 2 is for moderate bothersome/lasting 3-7 hours, 3 is for severely bothersome / lasted 7-24 hours, and 4 is for very severely bothersome / lasted > 24 hours. The severity and duration of symptoms are scored separately, which can not only analyse the overall state but also study the state of each item. The higher the score, the more serious the condition is.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | through study completion, an average of 3 months
  In a Numerical Rating Scale (NRS), patients are asked to select the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Beck Anxiety Inventory (BAI) | through study completion, an average of 3 months
  BAI measures anxiety severity through a self-statement manner. This scale contains 21 items with a four-point scoring method describing anxiety symptoms. On the scale, 0 is for "Not at All", 1 is for "Mildly but it did not bother me much", 2 is for "Moderately -it was not pleasant at times", and 3 is for "Severely - it bothered me a lot", to measure and infer the anxiety severity. Scores may range from 0 to 63 with 4 levels: minimal anxiety (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).

OTHER OUTCOMES:
TCM Body Constitution Scale Questionnaire | baseline, pre-intervention
  We will use the questionnaire developed by Prof. Wang Qi, School of Traditional Chinese Medicine, BUCM, to diagnose body constitution of subjects. There are totally 60 questions describing symptom of 9 constitutions, and each symptom is scored via 1-5: a score of one denotes that the symptom is not noticeable; while a score of five denotes that the symptom is severely bothersome.A score higher than 40% means that the patient belongs to that constitution.
TCM Syndrome Type Questionnaire | baseline, pre-intervention
  We will use a 16-item questionnaire to differentiate the type of dysmenorrhea. 16 questions describe symptoms of 5 syndrome type of dysmenorrhea, and each symptom is scored via 0-4: a score of zero denotes that the symptom is not noticeable; while a score of four denotes that the symptom is severely bothersome.A score higher than 75% means that the patient belongs to that syndrome type.
Tongue Image Features | through study completion, an average of 3 months
  We will distinguish the color of tongue with a color board, which used for judgement of TCM body constitution and syndrome type of dysmenorrhea

CONTACTS AND LOCATIONS:
Overall Officials: Shi Ping Zhang, Principal Investigator — Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine Building, Kowloon Tong, Kowloon, Hong Kong